CLINICAL TRIAL: NCT02314234
Title: Influence of Sugammadex on Facial Nerve Monitoring in Parotid Surgery
Brief Title: Improvement of Facial Nerve Monitoring in Parotid Surgery by Sugammadex
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, I-Cheng Lu, Visiting staff, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-20140248
Record Dates: First submitted 2014-12-04; First posted 2014-12-11 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Injury to Nerve During Surgery
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control group: did not receive muscle relaxant during anesthesia
- Sugammadex group: received single dose of rocuronium for anesthesia and sugammadex at skin incision
  Interventions: Drug: sugammadex (Bridion)

INTERVENTIONS:
Drug: sugammadex (Bridion) — single dose of sugammadex at skin incision
  Groups: Sugammadex group

SUMMARY:
To investigate the effectiveness of rapid reversal of rocuronium-induced neuromuscular block by sugammadex during IONM of facial nerve during parotid surgery

DETAILED DESCRIPTION:
Intraoperative neuromonitoring (IONM) of facial nerve has been applied in identifying and preserving facial nerve during parotid surgery. In this setting, even a single dose of nondepolarizing muscle relaxant may lead to delayed and weakened electromyography (EMG) signal in facial nerve monitoring during parotid surgery. The aim of this study was to investigate the effectiveness of rapid reversal of rocuronium-induced neuromuscular block by sugammadex during IONM of facial nerve during parotid surgery

ELIGIBILITY:
Inclusion Criteria:

* undergoing parotid surgery

Exclusion Criteria:

* facial nerve injury, renal failure, liver cirrhosis, neuromuscular disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient with facial nerve monitoring undergoing parotid surgery
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
evoked EMG amplitude of facial nerve | up to first post-op day

CONTACTS AND LOCATIONS:
Locations (1):
- I-Cheng Lu, Kaohsiung City, Taiwan